CLINICAL TRIAL: NCT03229733
Title: Design and Evaluation the Feasibility, Effects of Kinect-based Computer Games for Rehabilitation Training of Upper Extremity Function in Patients With Chronic Stroke
Brief Title: Design and Evaluation the Effects of Kinect-based Computer Games for U/E Training in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMRPG8E0931
Record Dates: First submitted 2017-07-23; First posted 2017-07-25 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2017-02

CONDITIONS: Stroke
Keywords: Stroke; Kinect; Rehabilitation; Upper limbs
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Patients randomized to the experimental group participate in exergames training with Kinect. The supervised OT chooses different games according to the patient's needs and abilities. During therapy patients are at sitting position. The game program will be adjusted when patients got improvement. After 30 minutes of exergames training, participants will receive a 30-minutes of traditional occupational therapy.
  Interventions: Device: Kinect; Behavioral: Traditional occupational therapy
- Control group (Active Comparator): Patients in the control group will receive individually tailored traditional occupational therapy consisting of the similar movement and dose as the experimental group doing by using the traditional equipment, such as climbing bar.
  Interventions: Behavioral: Traditional occupational therapy

INTERVENTIONS:
Device: Kinect — Receive Kinect games training for 30 minutes. There are 3 sections for 1 week; the intervention period will be 8 weeks
  Arms: Experimental group
Behavioral: Traditional occupational therapy — Patients will receive individually tailored conventional training consisting of the similar movement and dose by using the traditional equipment, such as climbing bar.

SUMMARY:
The aims of this study are to (i) develop exergames by using Kinect system for training UE function in patient with stroke; and (ii) to test the game's feasibility and effects in a group of patient with chronic stroke.

DETAILED DESCRIPTION:
Exercise based computer games can facilitate high volume complex task practice, enhance feedback of movement and increase motivation of participants. Those effects are difficult to achieve with standard rehabilitation therapy. The Kinect system is a camera-based controller which a player can use to directly control a game through body movement without the need for handheld controllers. Using Kinect to capture movement is a feasible way to help patients who have difficulties to hold controllers to play exergames. Scratch 2.0 is a programming language for kids from the MIT Media Laboratory. It is easy to use for game designing. Kinect2Scratch allows data from the Microsoft Kinect controller to be sent to Scratch, This means that game programs can be designed with motion control. The aims of this study were to i) develop exergames by using Scratch and Kinect system for training upper extremity function in patient with stroke; and ii) to test the game's feasibility and effects in a group of patient with chronic stroke.

This program will be done within two years. During the first year, investigators will design several exergames which are suitable for training upper extremity function in patient with stroke. Investigators will have several experts meetings, involved by physiatrists, occupational therapists and engineers to design the game. When a prototype game is created, investigators will invite two to four patients with stroke to pilot test the game. The game design will be completed till patients and therapists satisfy the design.

During the 2nd year, investigators will test the feasibility and effects of the exergames by doing a pilot randomized control trial. Investigators will recruit 60 patients with chronic stroke who are admitted to a rehabilitation ward for outpatient rehabilitation, and will randomize participants to experiment or control group. All participants will receive PT and OT training as routine. The additional intervention either exergames or conventional OT will be delivered for 8 weeks with 3 training sessions/week of up to 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* First ever ischemic or hemorrhagic stroke or former stroke without any significant residual motor impairment
* 3 months post stroke
* Impaired arm motor function at Brunnstrom stage 3-5
* Age 18 years or older

Exclusion Criteria:

* severe cognitive impairment defined as < 20 on Mini Mental State Examination
* visual disorders or neglect limiting the ability to comply with treatment regimen
* orthopedic problem or other neurological diagnosis that makes the UE dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Motor function assessed on Fugl-Meyer Assessment (FMA) | Change from baseline at 5 months
  The outcome will be measured at 3 time points: 0 week, 8 weeks, and 5 months after recruitment.

SECONDARY OUTCOMES:
The amount of movement assessed on Actigraph Assessment | Change from baseline at 2 months
  The outcome will be measured at 2 time points: 0 week, and 8 weeks after recruitment.
The upper extremity motor ability assessed on Wolf Motor Function Test (WMFT) | Change from baseline at 5 months
  The outcome will be measured at 3 time points: 0 week, 8 weeks, and 5 months after recruitment.
The quality of movement and amount of use assessed on Motor Activity Log (MAL) | Change from baseline at 5 months
  The outcome will be measured at 3 time points: 0 week, 8 weeks, and 5 months after recruitment.
The instrumental activities of daily living assessed on Nottingham Extended Activities of Daily Living Scale (NEADL) | Change from baseline at 5 months
  The outcome will be measured at 3 time points: 0 week, 8 weeks, and 5 months after recruitment.
The relevant for upper-extremity function self-report questionnaire on Stroke Impact Scale (SIS) | Change from baseline at 5 months
  The outcome will be measured at 3 time points: 0 week, 8 weeks, and 5 months after recruitment.
Standing balance assessed on The Functional reach test (FR) | Change from baseline at 5 months
  The outcome will be measured at 3 time points: 0 week, 8 weeks, and 5 months after recruitment.
Muscle power assessed on Medical Research Council Scale (MRC) | Change from baseline at 5 months
  The outcome will be measured at 3 time points: 0 week, 8 weeks, and 5 months after recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Wen Hung, Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Noorkoiv M, Rodgers H, Price CI. Accelerometer measurement of upper extremity movement after stroke: a systematic review of clinical studies. J Neuroeng Rehabil. 2014 Oct 9;11:144. doi: 10.1186/1743-0003-11-144. PMID 25297823
- [Result] Adams RJ, Lichter MD, Krepkovich ET, Ellington A, White M, Diamond PT. Assessing upper extremity motor function in practice of virtual activities of daily living. IEEE Trans Neural Syst Rehabil Eng. 2015 Mar;23(2):287-96. doi: 10.1109/TNSRE.2014.2360149. Epub 2014 Sep 24. PMID 25265612
- [Result] Wolf SL, Catlin PA, Ellis M, Archer AL, Morgan B, Piacentino A. Assessing Wolf motor function test as outcome measure for research in patients after stroke. Stroke. 2001 Jul;32(7):1635-9. doi: 10.1161/01.str.32.7.1635. PMID 11441212